CLINICAL TRIAL: NCT03992976
Title: Development of an Online, Interdisciplinary Intervention for Paediatric Chronic Pain Management
Brief Title: Development of an Online Program to Help Manage Chronic Pain in Children and Teenagers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 45429; 19BO01 (Other: Great Ormond Street Hospital for Children NHS Foundation Trust)
Record Dates: First submitted 2019-06-13; First posted 2019-06-20 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Paediatric Pain; Pain Management; Qualitative Research
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Teenagers with chronic pain: Semi-structured interviews followed by 'think-aloud' procedure in part two. Semi-structured interviews may last up to 1 hour and are audio-recorded. A pre-piloted interview schedule has been developed and will guide the conversation. 'Think-aloud' procedure involves showing participants some of the online content that has been developed on a computer screen, and asking them to say aloud their commentary on any aspects. Participants will be audio-recorded during the task, and it is not anticipated the task will take longer than 1 hour to complete. Each participant may only take part in one interview and one think-aloud procedure.
  Interventions: Other: Online Chronic Pain Management Intervention for Teenagers
- Parents of teenagers with chronic pain: Semi-structured interviews followed by 'think-aloud' procedure in part two. Semi-structured interviews may last up to 1 hour and are audio-recorded. A pre-piloted interview schedule has been developed and will guide the conversation. 'Think-aloud' procedure involves showing participants some of the online content that has been developed on a computer screen, and asking them to say aloud their commentary on any aspects. Participants will be audio-recorded during the task, and it is not anticipated the task will take longer than 1 hour to complete. Each participant may only take part in one interview and one think-aloud procedure.
  Interventions: Other: Online Chronic Pain Management Intervention for Teenagers

INTERVENTIONS:
Other: Online Chronic Pain Management Intervention for Teenagers — The intervention itself is currently under development. This development study is used to gather patient (teenager) insights, as well as insights from parents of these patients, which will inform the content and structure of the proposed intervention. This is done using qualitative-only techniques. Initial ideas for the intervention design mirror current clinical practices in paediatric chronic pain management. There are likely to be several different online modules, which include psychological techniques, medicine (advice), nursing (advice and guidance on non-pharmacological physical pain management), and physiotherapy (guidance for pacing and physiotherapy exercises). The intervention is intended to help teenagers employ a vast range of self-management techniques from these disciplines. Exact content is not yet refined as this is a development study.

SUMMARY:
This research seeks to develop an internet-based program to help teenagers manage pain at home using a variety of techniques from physiotherapy, medicine, psychology and nursing. This study uses interviews to investigate what content and features teenagers and their parents want to see in an online intervention for managing chronic pain in teenagers.

DETAILED DESCRIPTION:
This research seeks to develop an internet-based programme to help teenagers manage pain at home using a variety of techniques that mirror clinical practice. This includes content from medicine, physiotherapy, nursing and psychological techniques, such as relaxation.

The study will use interviews (one semi-structured interview and one 'think-aloud' interview per participant) to explore the question: What content and features do young people with chronic pain, and their parents want to see in an online pain management intervention?

The study seeks to recruit a group of teenagers from Great Ormond Street Hospital, as well as a group of parents. After the first round of interviews, participants have the option to be contacted about the second round.

Recruitment for the first round of interviews will continue up until the point where no additional insights are found by adding new data to the analysis ('point of saturation'). We anticipate 30 teenagers and 30 parents will be sufficient. We hope to recruit young people with a mixture of ages and sexes, as well as a mixture of different pain diagnoses, and parents with varying backgrounds and sexes where possible.

The insights gathered from this study will help develop a new program for managing chronic pain in teenagers, which we aim to make available through the NHS. The internet-based intervention hopes to contribute to successful chronic pain management at home, and may be used as an adjunct to clinical services, such as the Pain Control Service at Great Ormond Street Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12 to 17 years
* Adolescents experiencing chronic pain of any type (minimum duration of three months).
* Parents or legal guardians of adolescents, aged 12 to 17 years, who are experiencing chronic pain of any type (minimum duration of three months).

Exclusion Criteria:

* Unable to communicate in fluent, spoken English.
* Adolescents aged 18 years or over.
* Adolescents with chronic cancer pain that are continuing to undergo treatments to eradicate their primary cancer or have received these treatments in the last three months (maintenance therapies are acceptable).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Secondary care pain clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
8-item interview schedule | approximately 1 hour
  Patient-reported outcome collected from semi-structured interviews (dynamic measure). A pre-piloted interview schedule was developed for this specific study. The schedule contains questions about online pain management interventions for adolescents. There are 8 core questions, as well as a warm-up at the start and a debrief at the end.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Liossi, DPsych, Principal Investigator — University of Southampton, Great Ormond Street Hospital
Locations (1):
- University of Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised, transcribed data and audio-recordings will available via the University of Southampton file store for up to 10 years, in-line with university policy.

DOCUMENTS (1):
  • Study Protocol (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT03992976/Prot_000.pdf